CLINICAL TRIAL: NCT00666289
Title: Molecular Biology of Familial Myeloproliferative Disorders
Brief Title: Familial Myeloproliferative Disorders
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 07-0548-00105; P01CA108671-01A2 (NIH); MPD-RC 105 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia; Idiopathic Myelofibrosis
Keywords: polycythemia vera; essential thrombocythemia; idiopathic myelofibrosis; family clusters
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples from subjects and family members with myeloproliferative disease.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Myeloproliferative disorders occur in families, thus giving rise to the theory that it is a genetic disease that may be caused by an abnormal gene in the DNA that can be passed from one generation of family members to another. DNA can be gathered from family members through blood samples and the investigators will investigate (through DNA testing) to see if there are abnormal genes that may be responsible for causing the MPDs. Understanding which genes are responsible for causing MPDs can help develop ways to identify people who may be at risk for developing an MPD, allow for the development of better treatments, possibly a cure, or even prevent the development of MPDs.

ELIGIBILITY:
Inclusion Criteria:

* Families with 2 or more members diagnosed with polycythemia vera (PV), essential thrombocythemia (ET), PV and ET related myelofibrosis (PV-MF and ET-MF), idiopathic myelofibrosis (IM) or chronic myelogenous leukemia (CML).
* Healthy family members of subjects diagnosed with a myeloproliferative neoplasm (MPN).
* Participating subjects must be 7 years of age or older
* A written assent, parental permission or consent must be obtained prior to any study procedures being performed.

Exclusion Criteria:

* Subjects who have a known acquired cause of polycythemia (increased hemoglobin/hematocrit), such as people living in high altitudes (in excess of 14,000 feet), subjects with heart disease, left to right heart shunt, severe hypoxia, cyanotic congenital heart disease, or severe pulmonary disease, will be excluded from this study, secondary forms of thrombocytosis and secondary forms of myelofibrosis.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: families with multiple member diagnosed with myeloproliferative disease
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-03; Primary Completion 2015-01-20 (Actual); Study Completion 2015-06-20 (Actual)

PRIMARY OUTCOMES:
To determine a linkage from the DNA analyzed to find a gene that will allow for genetic evaluation of families with MPDs. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Josef Prachal, MD, Study Chair — Myeloproliferative Disorders-Research Consortium
Locations (6):
- United States (5):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Illinois at Chicago, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - Weill Cornell, New York, New York
  - University of Utah, Salt Lake City, Utah
- University of Florence, Florence, Italy